CLINICAL TRIAL: NCT04301908
Title: The Observational Cohort Study on Long-term Clinical Outcomes of Antiviral Therapy in Patients With Chronic Hepatitis B and Cirrhosis
Brief Title: A Cohort Study on Long-term Clinical Outcomes of Antiviral Therapy in Patients With Chronic Hepatitis B and Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of Hepatology Division 2, Beijing Ditan Hospital
Other Study IDs: DTXY024
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic hepatitis B; Interferon; Nucleoside (acid) analogs; HBV DNA; Hepatitis B surface antigen; Hepatocellular carcinoma
MeSH Terms: conditions — Hepatitis B, Chronic; Heartburn; Hepatitis B; Carcinoma, Hepatocellular | interventions — Interferons; Nucleosides; Acids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- antiviral therapy group: Patients with chronic hepatitis B and cirrhosis were treated with antiviral drugs
  Interventions: Drug: interferon

INTERVENTIONS:
Drug: interferon — Antiviral therapy for patients with chronic hepatitis B and cirrhosis. Antiviral therapies included interferon and / or nucleoside (acid) analogs, and patients who were continuously treated for more than 6 months were included in the study.
  Other Names: nucleoside (acid) analogues

SUMMARY:
This was a retrospective observational cohort study. The patients with chronic hepatitis B and cirrhosis who were treated with antiviral therapy in the Second Department of Liver Disease, Beijing Ditan Hospital, Capital Medical University from October 2008 to April 2020 were enrolled. Patients treated with antiviral drugs including interferon and/or nucleoside (acid) analogues lasting more than 6 months were included in the study. Interferon, nucleoside (acid) analogue monotherapy, combination therapy, sequential therapy, maintenance therapy and drug withdrawal therapy can all be included in the study. HBV DNA content, HBsAg/anti-HBs, HBeAg/anti-HBe, biochemical indexes, serum AFP and liver imaging (liver ultrasound) were collected before treatment (baseline), during treatment and after treatment. The virological response and clinical outcome after antiviral treatment for chronic hepatitis B were observed for at least 288 weeks, and the main evaluation indicators were the occurrence or reversal of cirrhosis complications, hepatocellular carcinoma and mortality. Secondary evaluation index: the influence factors of different clinical outcomes. To investigate the long-term virological response and clinical outcome of antiviral therapy in patients with chronic hepatitis B and liver cirrhosis and to clarify its influencing factors.

DETAILED DESCRIPTION:
This was a retrospective observational cohort study. The patients with chronic hepatitis B and cirrhosis who were treated with antiviral therapy in the Second Department of Liver Disease, Beijing Ditan Hospital, Capital Medical University from October 2008 to April 2020 were enrolled. Patients treated with antiviral drugs including interferon and/or nucleoside (acid) analogues lasting more than 6 months were included in the study. Interferon, nucleoside (acid) analogue monotherapy, combination therapy, sequential therapy, maintenance therapy and drug withdrawal therapy can all be included in the study. HBV DNA content, HBsAg/anti-HBs, HBeAg/anti-HBe, biochemical indexes, serum AFP and liver imaging (liver ultrasound) were collected before treatment (baseline), during treatment and after treatment. The virological response and clinical outcome after antiviral treatment for chronic hepatitis B were observed for at least 288 weeks, and the main evaluation indicators were the occurrence or reversal of cirrhosis complications, hepatocellular carcinoma and mortality. Secondary evaluation index: the influence factors of different clinical outcomes. To investigate the long-term virological response and clinical outcome of antiviral therapy in patients with chronic hepatitis B and liver cirrhosis and to clarify its influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75;
* Unlimited gender;
* Patients with chronic hepatitis B treated with interferon and / or nucleoside (acid) analogs (NA) antiviral therapy. All patients with chronic hepatitis B met the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015)
* No hormones and / or immunosuppressants and other hepatoprotective drugs;
* Sign a written informed consent.

Exclusion Criteria:

* Combined with other hepatitis virus (HCV, HDV) infections;
* Immune liver disease;
* HIV infection;
* long-term alcohol and / or other liver damage drugs;
* mental illness;
* Evidence of liver tumor (liver cancer or AFP> 100 ng / ml);
* Decompensated cirrhosis;
* Those who have serious heart, brain, lung, kidney and other system diseases that cannot participate in long-term follow-up;
* There are hormones and / or immunosuppressants and other hepatoprotective drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Antiviral therapy for patients with chronic hepatitis B and cirrhosis. Antiviral therapies included interferon and / or nucleoside (acid) analogs, and patients who were continuously treated for more than 6 months were included in the study. All patients with chronic hepatitis B and cirrhosis met the diagnostic criteria of China's Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
The rate of incidence or reversal of cirrhosis comorbidities, liver cancer, and the incidence of death | 288 weeks after antiviral therapy
  The incidence or reversal of cirrhosis comorbidities, the incidence of liver cancer, and the incidence of death

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No